CLINICAL TRIAL: NCT07319390
Title: Midpoint Transverse Process to Pleura Block vs Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Sleeve Gastrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU R226/2025
Record Dates: First submitted 2025-12-05; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Bariatric Sleeve Gastrectomy
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: data collector willnot know type of ths blick recieved
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (ESPB): Bilateral ESP (Active Comparator): block at T7 with 20 mL of 0.25% bupivacaine on each side
  Interventions: Procedure: Erector Spinae Plane Block (ESPB) group
- Group B (MTPB): Bilateral MTP (Active Comparator): block at T7 with 20 mL of 0.25% bupivacaine on each side
  Interventions: Procedure: Midpoint Transverse Process to Pleura Block (MTPPB)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESPB) group — will receive ESPB volume of 20 mls bupivacaine 0.25 % at level T7 bilaterally
  Arms: Group A (ESPB): Bilateral ESP
Procedure: Midpoint Transverse Process to Pleura Block (MTPPB) — will receive MTPB volume of 20 mls bupivacaine 0.25 % at level T7 bilaterally
  Arms: Group B (MTPB): Bilateral MTP

SUMMARY:
The aim of this study will be to compare between MTP and ESPB in terms of postoperative pain score in patients undergoing laparoscopic sleeve gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists (ASA) physical status II, of either sex Age ≥18 y.
* Undergoing laparoscopic sleeve gastrectomy
* BMI≥ 35

Exclusion Criteria:

* Patient refusal to give consent for the block
* Hypersensitivity to any of study medications
* Infection at site of the block
* Coagulopathy
* severe cardiac/hepatic/renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Mean postoperative pain numeric rating scale | pain will be evaluated first in postanesthesia care unit then at 1, 3, 6, 8, 12, 18, 24 hours posoperative
  Abdominal pain will be assessed using numeric rating scale which includes 10 degrees of which zero is no pain and 10 is maximum pain ever

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain Shams University hospitals, Cairo
  - Ain Shams university hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No